CLINICAL TRIAL: NCT02112825
Title: Exercise as an Adjunct Therapy to Reduce Blood Pressure in Chronic Kidney Disease
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1207M17821; R03DK097318 (NIH)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Focus Chronic Kidney Disease With Hypertension
Keywords: Exercise; blood pressure; chronic kidney disease
MeSH Terms: conditions — Motor Activity; Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): 12 weeks of blended supervised-home based exercise 3-4 times per week for 30-45 minutes
  Interventions: Behavioral: Exercise
- control (No Intervention): Control group asked to continue usual activities

INTERVENTIONS:
Behavioral: Exercise — Blended supervised-home based walking exercise 3-4 times per week for 30-45 minutes
  Arms: Exercise

SUMMARY:
The general objective of the study is to investigate the effect of regular aerobic exercise on resting and 24-hr blood pressure levels in men and women with stage 3-4 kidney disease and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* • Non-diabetic and >18 years of age

  * Diagnosed kidney disease with associated hypertension:
  * Non-nephrotic range proteinuria at diagnosis
  * No active glomerular disease or concomitant systemic inflammatory disease (e.g. lupus)
  * Systolic blood pressure >130 and/or diastolic blood pressure >80 mm Hg (on medication)
  * An estimated glomerular filtration rate of between 60 ml/min and 15 ml/min.
  * Individuals must be able to provide informed consent
  * Perform walking exercise training on a treadmill
  * Be able to participate in a 12-week supervised exercise program.

Exclusion Criteria:

* Currently participating in a formal exercise program
* Diabetes, active glomerular disease, or systemic inflammatory disease
* Requiring dialysis
* Have an Hematocrit <27%
* Uncontrolled hypertension (>200/110mmHg)
* Peripheral vascular disease.
* An inability to understand English or give consent. Other exclusion criteria are: any contraindications to exercise testing or training as indicated by the American College of Sports Medicine guidelines such as: Unstable coronary heart disease and symptomatic heart failure, exercise capacity limited by health problems such as angina, severe arthritis, or extreme dyspnea on exertion, progressive neuromuscular disease, pulmonary disease, or having undergone a coronary revascularization within the past 6 months prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
blood pressure | at week 0 and at week 12
  resting and 24-hour ambulatory blood pressure

SECONDARY OUTCOMES:
effective vascular compliance | at week 0 and at week 12
  Pulse wave velocity estimated systemic vascular resistance
endothelial function | at week 0 and at week 12
  measured by brachial artery flow mediated vasodilation
biomarkers associated with blood pressure | at week 0 and at week 12
  Circulating levels of angiotensin 2 Circulating levels of endothelin 1 asymmetric dimethylarginine

CONTACTS AND LOCATIONS:
Overall Officials: Ulf G Bronas, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States